CLINICAL TRIAL: NCT02982460
Title: The Effects of Isoinertial Training on Rotator Cuff Tendinopathy. A Randomized Controlled Double-blind Follow-up Trail. A Pilot Study
Brief Title: Effects of Isoinertial Training on Rotator Cuff Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UOMalaga
Record Dates: First submitted 2016-11-27; First posted 2016-12-05 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Rotator cuff tendinopathy; Eccentric exercise; Isoinertial training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isoinertial + eccentric exercise (Experimental): The isoinertial training will be based on 4 sets of 8 maximal repetitions using a YoYo-Squat (YoYo Technology AB, Stockholm, Sweden). This exercise device use the inertia of a spinning flywheel (moment inertia = 0.11 kg m-2), offering resistance during coupled concentric and eccentric actions, and allows for high demanding to rotator cuff exercises while offering the possibility to perform with an eccentric overload.Two initial repetitions in any set were aimed at accelerating the flywheel, before executing the subsequent 8 actions at maximal effort. Eccentric exercise will based on a set of 4 exercise implicating abduction, lateral rotation, extension and flexion of the shoulder.
  Interventions: Other: Isoinertial + eccentric exercise
- Eccentric exercise (Active Comparator): Eccentric exercise will based on a set of 4 exercise implicating abduction, lateral rotation, extension and flexion of the shoulder. Participants will attend three appointments per week over three weeks. They will complete three sets of 10 repetitions, with the exercises progressed in difficulty at each appointment.
  Interventions: Other: Eccentric exercise

INTERVENTIONS:
Other: Isoinertial + eccentric exercise — A session of isionertial + eccentric exercise covers the activity, strength and endurance of scapular muscles.
  Arms: Isoinertial + eccentric exercise
Other: Eccentric exercise — A session of eccentric exercise covers the strength of scapular muscles.
  Arms: Eccentric exercise

SUMMARY:
Rotator cuff tendinopathy (RCT) is regarded as a common and burdensome source of shoulder pain with prevalence estimated to be as high as 14% in general working-age population. RCT is a broad entity, including a vast variety of diagnosis such as shoulder impingement syndrome, RC tendinitis/tendinosis, as well as subacromial bursitis. The course of RCT is characterised by persistent pain and/or disability and/or recurrent episodes. It often leads to decrease function, lower health-related quality of life, poor sleep quality, work absenteeism, as well as patient's suffering. Previous studies support exercise as an adequate treatment in RCT. Nevertheless, our knowledge, there is no studies evaluating the effects of isoinertial training in RCT. Therefore, the aim of this study will be to pilot the methods proposed to conduct a substantive study to evaluate the efficacy of isoinertial training plus eccentric training versus eccentric training alone on improving pain and function in RCT. The objectives were to evaluate: (i) The process of recruitment and retention rates; (ii) Willingness of participants to be randomised; (iii) The extent of contamination between groups; (iv) Participant adherence with treatment. The secondary aim will be to analyse the effects of isoinertial training plus eccentric training versus eccentric training alone on rotator cuff strength, scapular muscle activity, and scapular muscle endurance in people with RCT.

DETAILED DESCRIPTION:
Study design and setting The design of the present study will be a randomized controlled single-blind trial with 2 follow-ups (one week and one month after intervention) that will be performed between January 2017 and March 2017 in one private physiotherapy clinic in Malaga, Spain. The outcomes will be assessed at baseline (t1), one week after intervention (t2), and one month after intervention (t3). Written informed consent will be acquired for all participants prior to their participation. The study will be implemented and reported in line with the CONSORT statement.

Recruitment Eligible participants who will be interested in the study will be asked to provide written informed consent to participate. Subsequently the patient-reported outcome measures will be completed to establish baseline pain, function, rotator cuff strength, scapular muscle activity, scapular muscle endurance and level of self-efficacy. After completion of the baseline measures, the participants will be randomly allocated to the isoinertial training plus eccentric or eccentric training groups. The measures of pain, function, rotator cuff strength, scapular muscle activity, scapular muscle endurance and self-efficacy will be repeated one week and one month after intervention. Anonymized age and gender will be collected for those participants who decline to take part in the study to assess the external validity of the recruited sample of participants. Participant data files will be stored in numerical order and in a secure and accessible place and manner. Participant files will be maintained in storage for a period of 3 years after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 years
* Willing and able to participate
* Primary complaint of shoulder pain
* No/minimal resting for shoulder pain
* Range of shoulder movement largely preserved
* Two out of three positive impingement tests: empty-can test, Hawkins-Kennedy test, modified Neer test
* Pain on isometric rotator cuff testing, usually abduction or lateral rotation.

Exclusion Criteria:

* Subjective feeling of instability and positive apprehension sign
* Positive scapular assistance and/or resistance test
* Partial or full ruptures of the rotator cuff
* Calcifications greater than 4 mm
* (Acromion type III (per Bigliani criteria)
* Bursitis
* History of shoulder fracture and/or shoulder surgery
* Glenohumeral disorders (inflammatory arthritis, osteoarthritis, osteonecrosis, cuff arthropathy, septic arthritis, adhesive capsulitis, glenohumeral instability); (viii) Regional disorders (cervical radiculopathy, brachial neuritis, nerve entrapment syndrome, sternoclavicular arthritis, reflex sympathetic dystrophy, and neoplasms)
* Systemic diseases
* Corticosteroid injection 3 months prior to the study treatment and within 1 months prior to the study treatment on other body parts.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
"Change from Baseline function at 1 month" | 1 month
  This outcome will be measured with the shoulder pain and disability index (SPADI)
"Change from Baseline pain at 1 month" | 1 month
  This outcome will be measured with the shoulder pain and disability index (SPADI)

SECONDARY OUTCOMES:
"Change from Baseline rotator cuff strength at 1 months" | 1 month
  The handheld dynamometer (HHD) (MicroFET 2, Hoggan Health Industries Inc., Biometrics, The Netherlands) was used to measure the following shoulder muscles strength: supraspinous, infraspinatus, subscapular, and teres minor.
"Change from Baseline scapular muscle activity at 1 months" | 1 month
  Surface electromyography (EMG; BTS FREEEMG 300, BTS S. p. A., Milan, Italy) was used to measure muscle activity. We attached an electrode to the supraspinous, infraspinatus, subscapular, and teres minor.
"Change from Baseline scapular muscle endurance at 1 months" | 1 month
  Endurance of the trapezius and serratus anterior muscles was assessed using the scapular muscle endurance (SME) test.
"Change from Baseline self-efficacy at 1 months" | 1 month
  Pain Self-Efficacy Questionnaire (PSEQ) contains 10 questions that will measure the patient's confidence in performing certain activities despite pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Luque Suarez, PhD, Principal Investigator — University of Malaga

IPD SHARING:
Plan to Share IPD: No